CLINICAL TRIAL: NCT00515203
Title: A Randomized, Double-Blind, Placebo-controlled Phase 1/2 Study to Determine the Safety and Efficacy of Romiplostim (AMG 531) in Thrombocytopenic Pediatric Subjects With Chronic Immune (Idiopathic) Thrombocytopenic Purpura
Brief Title: Safety and Efficacy Study of Romiplostim (AMG 531) to Treat ITP in Pediatric Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20060195
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Results first posted 2011-03-01 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Idiopathic Thrombocytopenic Purpura; Thrombocytopenia in Pediatric Subjects With Immune (Idiopathic) Thrombocytopenic Purpura (ITP); Thrombocytopenia in Subjects With Immune (Idiopathic) Thrombocytopenic Purpura (ITP)
Keywords: Immune (Idiopathic) Thrombocytopenic Purpura; Pediatric Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Purpura, Thrombocytopenic | interventions — romiplostim

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- II. (Placebo Comparator): 5 thrombocytopenic (as defined per protocol) subjects
  Interventions: Drug: Placebo
- I. (Experimental): 15 thrombocytopenic (as defined per protocol) subjects
  Interventions: Drug: AMG 531

INTERVENTIONS:
Drug: Placebo — Starting dose of 1.0 ug/kg. Dose adjustments are made throughout the study based on individual platelet counts.
  Arms: II.
Drug: AMG 531 — Starting dose of 1.0 ug/kg. Dose adjustments are made throughout the study based on individual platelet counts.
  Other Names: romiplostim
  Arms: I.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of romiplostim (AMG 531) in the treatment of thrombocytopenia in pediatric subjects with chronic ITP. We will also evaluate the efficacy of romiplostim (AMG 531) and characterize the pharmacokinetics of romiplostim (AMG 531). It is anticipated that romiplostim (AMG 531), when given at an effective dose and schedule, will be well tolerated treatment for thrombocytopenia among pediatric subjects with chronic ITP.

ELIGIBILITY:
Inclusion Criteria:

* Before any study-specific procedure, the appropriate written informed consent must be obtained. In addition to the written informed consent, the assent of the child from those subjects capable of providing assent must also be obtained if requested by the IRB/IEC.
* Diagnosis of ITP according to The American Society of Hematology (ASH) Guidelines at least six months prior to screening
* Age ≥ 12 months and < 18 years at enrollment
* The mean of two platelet counts taken during the screening period must be ≤ 30 x 10^9/L with no single count >35 x 10^9/L
* A serum creatinine concentration ≤ 1.5 times the laboratory normal range (for each age category)
* Adequate liver function; serum bilirubin ≤ 1.5 times the laboratory normal range
* Hemoglobin >10.0 g/dL

Exclusion Criteria:

* Known history of a bone marrow stem cell disorder (any abnormal bone marrow findings other than those typical of ITP must be approved by Amgen before a subject may be enrolled in the study)
* Known history of venous or arterial thrombotic or thromboembolic event
* Known history of congenital thrombocytopenia
* Known history of malignancy except basal cell carcinoma
* Known history of hepatitis B, hepatitis C, or HIV
* Known history of systemic lupus erythematosus, Evans Syndrome, or autoimmune neutropenia
* Known positive lupus anticoagulant or history of antiphospholipid antibody syndrome
* Known history of Disseminated Intravascular Coagulation, Hemolytic Uremic Syndrome, or Thrombotic Thrombocytopenic Purpura
* Currently receiving any treatment for ITP except for corticosteroids
* IV Ig or anti-D Ig within two weeks prior to the screening visit
* Rituximab (for any indication) within 14 weeks before the screening visit or anticipated use during the time of the proposed study
* Splenectomy within eight weeks of the screening visit
* Received hematopoietic growth factors including IL-11 (oprelvekin) within four weeks before the screening visit
* Received any alkylating agents within eight weeks before the screening visit or anticipated use during the time of the proposed study
* Subject is currently enrolled in or has not yet completed at least four weeks since ending other investigational device or drug trial(s), or subject is receiving investigational agent(s)
* Past or present participation in any study evaluating PEG-rHuMGDF, recombinant human thrombopoietin (rHuTPO), AMG 531, or related platelet product
* Pregnant (i.e. positive urine pregnancy test) or breast feeding
* Subject is not using adequate contraceptive precautions, if applicable.
* Known hypersensitivity to any recombinant E coli-derived product
* Subject has any kind of disorder that compromises the ability to comply with all study procedures

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Bussel JB, Buchanan GR, Nugent DJ, Gnarra DJ, Bomgaars LR, Blanchette VS, Wang YM, Nie K, Jun S. A randomized, double-blind study of romiplostim to determine its safety and efficacy in children with immune thrombocytopenia. Blood. 2011 Jul 7;118(1):28-36. doi: 10.1182/blood-2010-10-313908. Epub 2011 Apr 18. PMID 21502541
- [Background] Klaassen RJ, Mathias SD, Buchanan G, Bussel J, Deuson R, Young NL, Collier A, Bomgaars L, Blanchette V. Pilot study of the effect of romiplostim on child health-related quality of life (HRQoL) and parental burden in immune thrombocytopenia (ITP). Pediatr Blood Cancer. 2012 Mar;58(3):395-8. doi: 10.1002/pbc.23312. Epub 2011 Sep 9. PMID 21910213
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 19 Jul 2007 through 11 November 2008
Groups:
- Romiplostim: Romiplostim by subcutaneous injection once weekly at a starting dose of 1 µg/kg, adjusted based on weekly platelet counts to a maximum weekly dose of 10 µg/kg
- Placebo: Placebo by subcutaneous injection once weekly
Period: Overall Study
Arm/Group | Romiplostim | Placebo
Started | 17 | 5
Completed | 17 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Romiplostim | Placebo | Total
Number analyzed (Participants) | 17 | 5 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.4 (5.4) | 9.8 (4.6) | 9.5 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 13 | 3 | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 9 | 4 | 13
  Black or African American | 5 | 0 | 5
  Hispanic or Latino | 3 | 0 | 3
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Weeks With Platelet Count ≥ 50 x 10^9/L
Description: The number of weeks with platelet count ≥ 50 x 10^9/L during the 12 week treatment period.
Time Frame: 12-week treatment period
Population: Efficacy Analysis Set, composed of all randomized participants
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 17 | 5
Weeks | 5.65 (3.00) | 0.00 (0.00)
Statistical Analysis 1: Comparison: Romiplostim vs Placebo; Test type: Superiority or Other; p = 0.0019, Cochran-Mantel-Haenszel

2. Secondary Outcome: Bleeding Events (Grade 2 or Higher)
Description: Total number of bleeding events (Grade 2 or higher, i.e., mild to life-threatening, as defined in the protocol) for each participant during Weeks 2-13 (end-of-study visit for non-responders)
Time Frame: 12-week treatment period (Weeks 2 - 13)
Population: Efficacy Analysis Set, composed of all randomized participants
Measure: Mean (Standard Deviation); unit: Events per participant
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 17 | 5
Events per participant | 0.41 (1.00) | 0.00 (0.00)
Statistical Analysis 1: Comparison: Romiplostim vs Placebo; Test type: Superiority or Other; p = 0.3651, Cochran-Mantel-Haenszel

3. Secondary Outcome: Platelet Count ≥ 50 x 10^9/L for Two Consecutive Weeks
Description: Participant incidence of achieving a platelet count ≥50 x 10^9/L for two consecutive weeks during the 12 week treatment period.
Time Frame: 12-week treatment period
Population: Efficacy Analysis Set, composed of all randomized participants
Measure: Number; unit: Participants
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 17 | 5
Participants | 15 | 0
Statistical Analysis 1: Comparison: Romiplostim vs Placebo; Test type: Superiority or Other; p = 0.0008, Fisher Exact

4. Secondary Outcome: Increase in Platelet Count ≥ 20 x 10^9/L Above Baseline for Two Consecutive Weeks
Description: Participant incidence of achieving an increase in platelet count ≥20 x 10^9/L above baseline for two consecutive weeks during the 12 week treatment period.
Time Frame: 12-week treatment period
Population: Efficacy Analysis Set, composed of all randomized participants
Measure: Number; unit: Participants
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 17 | 5
Participants | 15 | 0
Statistical Analysis 1: Comparison: Romiplostim vs Placebo; Test type: Superiority or Other; p = 0.0008, Fisher Exact

5. Secondary Outcome: Requirement for Rescue Therapy (as Defined Per Protocol)
Description: Participant required rescue therapy (as defined per protocol) during the 12 week treatment period.
Time Frame: 12-week treatment period
Population: Efficacy Analysis Set, composed of all randomized participants
Measure: Number; unit: Participants
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 17 | 5
Participants | 2 | 2
Statistical Analysis 1: Comparison: Romiplostim vs Placebo; Test type: Superiority or Other; p = 0.2098, Fisher Exact

6. Primary Outcome: Adverse Events
Description: Occurrence of one or more adverse events in the participant during the 12-week treatment period
Time Frame: 12 weeks
Population: Safety Analysis Set, composed of all participants who received at least one dose of study medication
Measure: Number; unit: Participants
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 17 | 5
Participants | 16 | 5

ADVERSE EVENTS:
Time Frame: 12 week treatment period
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Placebo | Romiplostim
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/17
Other Adverse Events (participants affected / at risk) | 5/5 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | Romiplostim (N=17)
Influenza (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | Romiplostim (N=17)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Chapped lips (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Chest discomfort (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 4
Hypersensitivity (Immune system disorders) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2
Otitis media (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Spleen palpable (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 6
Emotional disorder (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Urethral disorder (Renal and urinary disorders) | 0 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.